CLINICAL TRIAL: NCT01880606
Title: Probe-based Confocal Laser Endomicroscopy in Colonoscopic Surveillance of Patients With Primary Slerosing Cholangitis Related Inflammatory Bowel Disease (PSC-IBD)
Brief Title: Endomicroscopy in Primary Sclerosing Cholangitis Related Inflammatory Bowel Disease Surveillance
Acronym: pCLE-PSC-IBD
Status: Completed | Type: Observational
Sponsor: Karolinska University Hospital (Other)
Responsible Party: Principal Investigator, Aldona Dlugosz, MD, PhD consultant, Karolinska University Hospital
Other Study IDs: PSC-IBD2012
Record Dates: First submitted 2013-06-12; First posted 2013-06-19 (Estimated); Last update posted 2015-04-27 (Estimated); Status verified 2015-04

CONDITIONS: Primary Sclerosing Cholangitis; Inflammatory Bowel Disease
MeSH Terms: conditions — Cholangitis, Sclerosing; Inflammatory Bowel Diseases | interventions — Colonoscopy

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Biospecimen Retention: Samples With DNA — whole blood, serum, tissue
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- patients with PSC-IBD: Only patients, colonoscopy with endomicroscopy
  Interventions: Procedure: colonoscopy with endomicroscopy

INTERVENTIONS:
Procedure: colonoscopy with endomicroscopy — Examination will be performed in two steps. On the way from rectum to caecum, mucosa will be evaluated with white light endoscopy and random biopsies will be taken according to the routine standard with minimum of 2 biopsies from each 10 cm of colon. On the way back (from caecum to rectum) mucosa will be stained with indigo carmine and after intravenous fluorescein injection all macroscopically abnormal lesions will be examined by endomicroscopy and biopsied. Additionally, all places where random biopsies were taken will be also examined with endomicrosopy.

SUMMARY:
Evaluation of the efficacy of laser-based endomicroscopy as a complement to white-light colonoscopy and chromoendoscopy for early detection of colon dysplasia in patients with PSC-IBD. White-light colonoscopy is a routinely used procedure in colorectal cancer surveillance programs. However, it does not permit detection of early dysplastic lesions. Chromoendoscopy by applying a dye (indigo-carmine) through the colonoscope helps to identify flat lesions but is not suitable for accurate endoscopic diagnosis of dysplasia and intraepithelial neoplasia Under this aim we will perform a clinical study evaluating a newly developed technique allowing for in vivo confocal microscopy assessment of the colon mucosa using laser-based endomicroscopy together with intravenous administration of fluorescein (FITC).

DETAILED DESCRIPTION:
Chromoendoscopy by applying a dye (indigo-carmine) through the colonoscop is the new standard for cancer surveillance in patients with IBD . It gives the opportunity to identify suspected areas of dysplasia and to take targeted biopsies. The diagnostic accuracy improves and the chances for detecting dysplastic areas increase. In recent years new endoscopic techniques have been developed, including laser-based endomicroscopy. There is an increasing need for structured evaluation of the efficiency of these techniques. Laser-based endomicroscopy, taking in vivo confocal microscopy pictures during the colonoscopy examination, is the most promising new method. This method is established in highly rated centers for the early diagnosis of neoplasia in the bile ducts and the esophagus but its role for detection early malignancies in the colon is not known and studying this issue is of very high clinical value.

Specific questions: Does the use of laser-based endomicroscopy increase the chances for early detection of dysplasia? What is the intraobserver variability? What is the learning curve for interpretation of confocal microscopy pictures? Material and methods: A laser-based endomicroscope (Cellvizio®, Mauna Kea Technologies) have been acquired and the examination procedure has been established at the Unit for Gastroenterology and Hepatology, Karolinska University Hospital Huddinge. Eighty patients with PSC and IBD included in annual surveillance with colonoscopy with routine biopsy regime will be included in the study. After informed consent, patients are investigated with laser-based endomicroscopy during surveillance colonoscopy. Each colonic segment will be examined before and after staining with indigo-carmin. After intra-venous fluorescein (FITC) injection, all macroscopically abnormal lesions will be examined by endomicroscopy. Intravenous administration of FITC makes it possible to obtain in vivo microscopic pictures with up to a 1000x magnification of the colon mucosa. The Cellvizio® technique allows for evaluation of epithelial and endothelial cell structures in areas with suspicious changes as well as for acquisition of directed biopsies. Confocal pictures from all sites where biopsies have been taken are saved for future blind re-evaluation. The biopsies are taken according to the routine standard with minimum of 2 biopsies from each 10 cm in the colon. For the immunological and microbiological (specific aim 2) parts of the study, additional 16 biopsies are gathered from left, transverse, and right colon. All the laser-based endomicroscopy pictures and sequences are saved for further evaluation and further application in arranging pedagogical sessions for evaluation of the learning curve of the technique.

ELIGIBILITY:
Inclusion Criteria:

* clinical diagnosis of PSC-IBD

Exclusion Criteria:

* the lack of informed consent, allergy to fluorescein, B-blockers treatment

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Eighty patients with PSC and IBD included in annual surveillance with colonoscopy with routine biopsy regime will be included in the study.
Sampling Method: Probability Sample
Enrollment: 69 (Actual)
Dates: Start 2011-08; Primary Completion 2013-12 (Actual); Study Completion 2014-06 (Actual)

PRIMARY OUTCOMES:
Sensitivity and specificity of endomicroscopy versus white light endoscopy in detection of dysplastic lesions in colon using histological assesment as a gold standard. | one year

SECONDARY OUTCOMES:
measurement of number of dysplastic lesions discovered by adding pCLE to white-light endoscopy | one year

CONTACTS AND LOCATIONS:
Overall Officials: Annika Bergquist, PhD, Study Chair — Gastro Center Karolinska Institute
Locations (1):
- Gastro Center Karolinska University Hospital, Stockholm, Sweden